CLINICAL TRIAL: NCT02667171
Title: COPD Online Rehabilitation (CORe) - a Randomized, Multicenter Telemedicine Intervention Study
Brief Title: COPD Online Rehabilitation (CORe)
Acronym: CORe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: TrygFonden, Denmark (Industry); Danish Lung Association (Other); Region Capital Denmark (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Henrik Hansen, Ph.D. student, Physiotherapist, Master of Health Sciences, Project Manager,, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-12910 01-01-01
Record Dates: First submitted 2016-01-12; First posted 2016-01-28 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled, assessor- and statistician blinded, superiority, multicentre trial with two parallel-groups. Online COPD Rehab versus Coventional COPD rehab
Who Masked: Investigator, Outcomes Assessor
Masking Description: All assessors are blinded to group allocation and previous test results. Due to the nature of the study the patients cannot be blinded, but prior to the assessments they are reminded not to disclose their group allocation to the assessors. In case of failure keeping the outcome assessor blinded (that is, if a participant reveals his/her allocation) a second assessor will be available to step in and conduct the assessment on another day.
  To avoid investigators (subconscious) bias the biostatistician who perform the data analyses and validate the results will be blinded to group allocation.
  The research group will interpret the results, and the conclusion will be prepared in two versions before the allocation code is broken (one assuming that arm A is the intervention, and one assuming that arm B is the intervention).
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Active Comparator): The control group will receive standardized conventional supervised COPD rehabilitation, delivered in groups. Rehabilitation contains exercise training and education sessions twice a week for a duration of 8-12 weeks.
  Interventions: Behavioral: Supervised COPD Rehabilitation (control group)
- Online COPD rehabilitation (Experimental): Supervised Online COPD rehabilitation, delivered in groups through a computer screen in patients own home. Rehabilitation contains exercise training and education sessions three times per week for a duration of 10 weeks.
  Interventions: Behavioral: Online COPD rehabilitation (experimental)

INTERVENTIONS:
Behavioral: Supervised COPD Rehabilitation (control group) — The control group receives standardized conventional supervised COPD rehabilitation (CCR) in groups. Rehabilitation contains exercise training and education sessions twice a week for a duration of 8-12 weeks. The CCR will last 60-120 minutes each session (50% exercise and 50% education).
  Physical Exercises in CCR consist endurance based at Borg dyspnea 4-7 for 20-30 minutes and resistance training for upper and lower limb at 50-80% of one repetition maximum of 2-3 sets. Educations sessions consist information a dialogue regarding, life with COPD, participants topics, Medication, daily activity, Nutrition, Smoking cessation, Respiratory and relaxation exercises.
  Arms: Control group
Behavioral: Online COPD rehabilitation (experimental) — Supervised Online COPD rehabilitation, delivered in groups through a computer screen in patients own home. Rehabilitation contains exercise training and education sessions three times per week for a duration of 10 weeks. Each session lasts for 60minutes (60% exercise 40% education). Physical exercises consist high repetitive time-based muscle endurance training, including 5-7 upper and lower limb exercises, performed with a volume of four sets per exercise equivalent to 50-80% of one repetition. Self-rated Borg CR-10 score equivalent from moderate to very strong shortness of breath in active phases.
  Educations consists same information as for the control group.
  Arms: Online COPD rehabilitation

SUMMARY:
International and national publications emphasize that COPD rehabilitation is a key cornerstone in the standard treatment of COPD, based on more than 15 years of research in COPD rehabilitation. COPD rehabilitation improves quality of life, anxiety and depression and physical function. COPD rehabilitation including special physical training, patient-directed education and smoking cessation is core rehabilitation elements, which today are recommended as mandatory content in standard COPD rehabilitation.

Standard COPD rehabilitation is an established offer in all regions and municipalities in Denmark. It is however a well-known challenge, that persons with the most severe COPD symptoms and co-morbidities are most likely not to receive COPD rehabilitation. Frequent exacerbations, socially isolation, transport distance to rehabilitation are main reasons why people with severe COPD disease deliberately chooses not to receive COPD rehabilitation. Why there at present are no rehabilitation alternatives for patients with the most severe COPD symptoms, supervised COPD Online rehabilitation in groups, delivered by health professionals in the COPD patients' own home via a computer screen could likely encourage more people to participate. The number of RCT's investigating the effect of supervised Online delivered COPD rehabilitation in groups versus established COPD rehabilitation are very limited.

The purpose of this randomized study is to investigate the short-term and long-term efficacy of 10 weeks of online COPD rehabilitation versus conventional supervised COPD rehabilitation in people with severe and very severe COPD. The outcome of the intervention is measured on walking distance, muscle endurance, activity level, quality of life and COPD symptoms respectively. Outcomes are measures before intervention start, end of intervention. This study also collects follow-up update after 3, 6 and 12 month. The follow-up data will be in separate publication.

Hypothesis

1. COPD online rehabilitation provides significant larger improvements than the usual care on walking distance, muscle endurance, activity level, and quality of life and COPD symptoms in people with severe and very severe COPD.
2. COPD online rehabilitation and conventional COPD rehabilitation, provides clinically relevant improvement on walking distance, muscle endurance, activity level, quality of life and COPD symptoms in people with severe and very severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD defined as a ratio of forced expiratory volume at one second (FEV1) to forced vital capacity < 0.70
* FEV1 <50%, corresponding to severe or very severe COPD
* Symptoms equivalent to the Medical Research Council (MRC) from 2 to 5

Exclusion Criteria:

* Concurrent participation in or recent completion of pulmonary rehabilitation within the last six months.
* Dementia/ Cognitive impairment or uncontrolled psychiatric illness,
* An impaired hearing and / or vision which causes the instructions in the rehabilitation is not understood.
* Unable to understand and / or speak Danish.
* Unable to read Danish.
* Severe co-morbidity that are contraindicated to rhe clinical exercise protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in 6-Minute Walk Test Distance (6MWT) | baseline (before intervention), after 10 weeks, after 22 weeks (average of 3 month follow up)
  In-clinic test that measures exercise capacity

SECONDARY OUTCOMES:
Change in 30 second sit-to-stand test (30-STST) | baseline (before intervention), after 10 weeks, after 22 weeks (average of 3 month follow up)
  In-clinic test that measures muscle endurance/strength
Change in Activity level (ActivPAL) | Worn by the patients around the clock for 5 days in a private home at baseline (before intervention), after 10 weeks, after 22 weeks (average of 3 month follow up)
  Worn by the patients around the clock for 5 days in a private home.
Change in Clinical COPD Questionaire (CCQ) | baseline (before intervention), after 10 weeks, after 22 weeks (average of 3 month follow up)
  Patient completed questionnaires that assess quality of life and COPD symptoms. Ten Item questionaire with total score from 0-60 points.
Change in COPD Assessment Test (CAT) | baseline (before intervention), after 10 weeks, after 22 weeks (average of 3 month follow up)
  Patient completed questionnaires that assess quality of life and COPD symptoms. Five item questionaire with total score from 0-40 points.
Change in Hospital Anxiety and Depression Scale (HADS) | baseline (before intervention), after 10 weeks, after 22 weeks (average of 3 month follow up)
  Patient completed questionnaires that assess anxiety and depression symptoms. Seven item domain questions for depression with total score form 0-21 point. Seven item domain questions for anxiety with total score fra 0-21 points. Total score from 0-42 points
Change in Euro Qol (EQ5D) | baseline (before intervention), after 10 weeks, after 22 weeks (average of 3 month follow up)
  Patient completed questionnaires that assess quality of life. Total score fra 0-1 on EQ5D-health domain. Total score from 0-100mm on EQ5D-vas domain. No total domain score
Total attendance in rehabilitation | after 10 weeks
  registered
number of hospital admissions | number of hospital admissions - after 10 weeks, after 22 weeks (average of 3 month follow up), after 36 weeks (average of 6 month follow up), after 62 weeks (average of 12 month follow up)
  from registers
Number of hospital days | number of hospital days - after 10 weeks, after 22 weeks (average of 3 month follow up), after 36 weeks (average of 6 month follow up), after 62 weeks (average of 12 month follow up)
  from registers
Outpatient visits in hospital and at general practioner | number of outpatients visits in hospital and at general practioner - after 10 weeks, after 22 weeks (average of 3 month follow up), after 36 weeks (average of 6 month follow up), after 62 weeks (average of 12 month follow up)
  from registers
Mortality | after 10 weeks, after 22 weeks (average of 3 month follow up), after 36 weeks (average of 6 month follow up), after 62 weeks (average of 12 month follow up)
  from registers

CONTACTS AND LOCATIONS:
Overall Officials: Anne Frølich, MD, PhD, Study Chair — Research Unit for Chronic Diseases and Telemedicine
Locations (7):
- Denmark (7):
  - Bispebjerg and Frederiksberg Hospital, Copenhagen, Copenhagen Northwest
  - Amager Hospital, Copenhagen
  - Frederikssund hospital, Frederikssund
  - Gentofte Hospital, Hellerup
  - Herlev Hospital, Herlev
  - Hillerød hospital, Hillerød
  - Hvidovre Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. Data sharing plan: Supervised pulmonary tele-rehabilitation versus pulmonary rehabilitation in severe COPD: a randomised multicentre trial. When and for how long the data will become/be available? Data available until 31 December 2021. Proposal for data use should be addressed to henrik. hansen. 09@ regionh. dk. Data access in Denmark are under very strict juristic data protection law. Any possible access or sharing demands a part application to; (1) Danish Data Protection Agency, (2) Ethics Committee of the Capital Region, (3) National Health Data Authorities.
  Only if the applications are approved data will be considered available for sharing.
  The authors will not be able to support this process and a prolonged process must be expected.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 31st of December 2021
Access Criteria: please res plan description above

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633
- [Derived] Hansen H, Bieler T, Beyer N, Kallemose T, Wilcke JT, Ostergaard LM, Frost Andeassen H, Martinez G, Lavesen M, Frolich A, Godtfredsen NS. Supervised pulmonary tele-rehabilitation versus pulmonary rehabilitation in severe COPD: a randomised multicentre trial. Thorax. 2020 May;75(5):413-421. doi: 10.1136/thoraxjnl-2019-214246. Epub 2020 Mar 30. PMID 32229541
- [Derived] Hansen H, Bieler T, Beyer N, Godtfredsen N, Kallemose T, Frolich A. COPD online-rehabilitation versus conventional COPD rehabilitation - rationale and design for a multicenter randomized controlled trial study protocol (CORe trial). BMC Pulm Med. 2017 Nov 16;17(1):140. doi: 10.1186/s12890-017-0488-1. PMID 29145831